CLINICAL TRIAL: NCT02419040
Title: Treatment of Calcific Tendinitis of the Rotator Cuff - a Multi-centre, Randomized and Sham Controlled Trial (KALK Study)
Brief Title: Treatment of Calcific Tendinitis of the Rotator Cuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Helse Fonna (Other); Oslo University Hospital (Other); Sykehuset i Vestfold HF (Other); Haraldsplass Deaconess Hospital (Other); University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Stefan Moosmayer, MD, PhD, Vestre Viken Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KALK-001
Record Dates: First submitted 2015-04-10; First posted 2015-04-17 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Pain; Tendonitis; Calcinosis; Shoulder Impingement Syndrome
Keywords: shoulder pain; rotator cuff; calcific tendonitis; barbotage
MeSH Terms: conditions — Shoulder Pain; Tendinopathy; Calcinosis; Shoulder Impingement Syndrome | interventions — Adrenal Cortex Hormones; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Barbotage (Experimental): Ultrasound guided needling, lavage and steroid/lidocain injection (20 mg Triamcinolon/9 ml Lidocain 1%) Ultrasound guided lidocain injection (10 ml Lidocain 1%, sham group) and home exercises
  Interventions: Procedure: Barbotage
- Corticosteroid injection (Active Comparator): Ultrasound guided steroid/lidocain injection (20 mg Triamcinolon/9 ml Lidocain 1%) and home exercises
  Interventions: Procedure: Corticosteroid injection
- Lidocain injection (sham) (Sham Comparator): Ultrasound guided lidocain injection (10 ml Lidocain 1%, sham group) and home exercises
  Interventions: Procedure: Lidocain injection (sham)

INTERVENTIONS:
Procedure: Barbotage — A 18-gauge needle connected to a 5 ml syringe with 4 ml of saline solution will be used to puncture the calcification with freehand technique and under constant sonographic monitoring. With the tip of the needle placed in the center of the deposit, the calcification will be flushed. Finally, a new 21-gauge needle will be introduced into the subacromial-subdeltoid bursa and 9 ml of 1% Lidocain hydrochlorid and 1 ml (20 mg) of Triamcinolon will be injected into the subacromial-subdeltoid bursa. All patients will be instructed by a physioteherapist in home exercises.
  Other Names: 20 mg Triamcinolon/; 9 ml Lidocain 1%
  Arms: Barbotage
Procedure: Corticosteroid injection — The tip of the 18-gauge needle will be placed in the soft parts outside of the rotator cuff and movements mimicking the lavage procedure will be performed. A lavage procedure usually takes 5 minutes and the same period of time will have to be used for the mimicking maneuver. Finally, a new 21-gauge needle will be introduced into the subacromial-subdeltoid bursa and 9 ml of 1% Lidocain hydrochlorid and 1 ml (20 mg) of Triamcinolon will be injected into the subacromial-subdeltoid bursa. All patients will be instructed by a physioteherapist in home exercises.
  Other Names: 9 ml Lidocain 1%; 20 mg Triamcinolon/
  Arms: Corticosteroid injection
Procedure: Lidocain injection (sham) — The tip of the 18-gauge needle will be placed in the soft parts outside of the rotator cuff and movements mimicking the lavage procedure will be performed. A lavage procedure usually takes 5 minutes and the same period of time will have to be used for the mimicking maneuver. Finally, a new 21-gauge needle will be introduced into the subacromial-subdeltoid bursa and 10 ml of 1% Lidocain hydrochlorid will be injected into the subacromial-subdeltoid bursa. All patients will be instructed by a physioteherapist in home exercises.
  Other Names: 9 ml Lidocain 1%
  Arms: Lidocain injection (sham)

SUMMARY:
The purpose of this study is to determine whether the combination of removal of the calcification in calcific tendinitis of the shoulder (supraspinatus and/or infraspinatus tendon) by aspiration with a needle and syringe (barbotage) and a corticosteroid injection is more effective than corticosteroid or sham injection alone.

DETAILED DESCRIPTION:
Barbotage is a sonographically guided percutaneous needle aspiration and lavage of the calcium deposit in calcific tendinitis of the shoulder. Persisting pain in cacific tendinitis is considered to be a consequence of increased tendon volume or changed tendon texture in the area of the calcification which leads to secondary impingement and inflammation. Consequently, removal of the deposit should be a causal treatment measure.

Scientific evidence for the efficacy of the barbotage procedure in patients with persistent symptoms from calcific tendinitis is still limited. The cyclic often self-limiting course of the disease, and an anticipated placebo effect, questions about the method's efficacy can only be answered by high-quality randomized studies. In this trial the investigators want to randomize a cohort of patients to (1) Ultrasound guided needling, lavage and subacromial steroid injection, (2) Ultrasound guided subacromial steroid injection or (3) Ultrasound guided lidocain injection (sham). The investigators want to follow the patients over two years with repeated testing with a set of validated outcome measures together with radiologic re-examinations. The investigators want to find out whether the active treatments (1, 2) are more effective than the sham treatment and whether there are differences in outcome between the two active treatments. To increase the generalizability of the investigators' results, the investigators want to perform the study as a multi-centre study.

ELIGIBILITY:
Inclusion Criteria:

1. 30 years or older
2. 3 months or more of shoulder pain
3. Moderate to strong pain localized on the top and/or lateral side of the shoulder, exaggerated by activities above shoulder level
4. Painful arc
5. Positive Hawkin's test and/or Neer's sign for impingement
6. Finding of one or more calcifications ≥5 mm in size on a standard anteriorposterior radiograph, localized proximally to the greater tubercle, together with a sonographic finding of one or more calcifications ≥5 mm in size on the short or long axis view, localized in the supraspinatus or infraspinatus tendon
7. Morphological radiographic appearance of Molé type A, B or C12 (appendix 2) A: Dense, homogeneous with well-defined limits B: Dense, fragmented with well-defined limits C: Heterogeneous with poorly defined limits and sometimes with a punctuate appearance
8. Ability to understand written and spoken Norwegian (Swedish/English)
9. Existing signed informed consent and expected cooperation of the patients for the treatment and the follow-up

Exclusion criteria:

1. Clinical and radiological signs of a recent spontaneous release of the deposit such as a sudden change in size or density of the deposit on ultrasound together with an acute onset of extreme shoulder pain
2. Clinical signs of shoulder instability, glenohumeral arthritis, AC pathology, inflammatory arthropathy, fibromyalgia, frozen shoulder or cervical radiculopathy
3. Sonographic signs for a rotator cuff tear (full thickness or partial thickness) and of a tear or a dislocation of the long head of the biceps tendon
4. A history of surgical treatment of the relevant shoulder
5. A subacromial injection with a corticosteroid during the last 3 months before inclusion
6. Medical contraindications for any of the invasive procedures
7. One of the following contraindications for the use of Lidocaine 10 mg/ml: Patients with serious hypovolaemia, known cardiac conduction disturbances, epilepsy or porphyrias, patients with known serious dysfunction of the liver or the kidneys.
8. One of the following contraindications for the use of Triamcinolone 20 mg/ml: Patients with systemic infections unless specific anti-infective therapy is employed, patients with a local infection in the area of application, patients recently vaccinated with live vaccines, patients with known diabetes mellitus, renal or cardiac insufficiency, ulcerating colitis, gastric ulcer, psychosis, idiopathic thrombocytopenic purpura, or ocular herpes simplex.
9. Concomitant medication with one of the following medicinal products: Anti-arrythmics such as mexiletine or class III antiarrythmics (e.g. amiodarone), muscle relaxants (e.g. suxamethonium) or antipsychotics (e.g. pimozide, sertindole, olanzapine, quetiapine, zotepine, tropisetrone, dolasetron), antibiotics such as quinopristin/dalfopristin.
10. Any history of prior allergic/hypersensitivity reactions related to the study medication
11. Knowledge of an ongoing pregnancy (Fertile women not using contraception and who are uncertain whether they are pregnant or not will have to perform a pregnancy test)
12. Nursing women

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 4 months
  Shoulder pain and disability

SECONDARY OUTCOMES:
Oxford Shoulder Score | after 2 and 6 weeks, and 8, 12 and 24 months
  Shoulder pain and disability
QuickDASH Disability of shoulder, arm and hand | after 2 and 6 weeks, and 4, 8, 12 and 24 months
  Shoulder pain and disability
EQ 5D-5L | 4, 8, 12 and 24 months
  Health related quality of life
Cross-over of patients | 4, 8, 12 and 24 months
  number of patients crossing over to other group or other treatment
Adverse-events | 2 and 6 weeks, and 4 months
  Patient reported adverse events

OTHER OUTCOMES:
Size of calcific deposits | 4 and 24 months
  Measured in millimeter AP radiographs
Volume of removed calcific deposit | Baseline
  Volume of removed calcific deposit in milliliter

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Moosmayer, MD, PhD, Principal Investigator — MHH Martine Hansens Hospital
Locations (1):
- Martina Hansen's Hospital, Sandvika, Norway

REFERENCES:
- [Background] Moosmayer S, Ekeberg OM, Hallgren HB, Heier I, Kvalheim S, Blomquist J, Pripp AH, Juel NG, Kjellevold SH, Brox JI; KALK study group. KALK study: ultrasound guided needling and lavage (barbotage) with steroid injection versus sham barbotage with and without steroid injection - protocol for a randomized, double-blinded, controlled, multicenter study. BMC Musculoskelet Disord. 2017 Apr 4;18(1):138. doi: 10.1186/s12891-017-1501-9. PMID 28376756
- [Background] Robinson DM, McInnis KC, Rhim HC, Tsitsilianos N. Lavage treatments for calcific rotator cuff tendinopathy. BMJ. 2023 Oct 11;383:2248. doi: 10.1136/bmj.p2248. No abstract available. PMID 37821118
- [Result] Moosmayer S, Ekeberg OM, Hallgren HB, Heier I, Kvalheim S, Juel NG, Blomquist J, Pripp AH, Brox JI. Ultrasound guided lavage with corticosteroid injection versus sham lavage with and without corticosteroid injection for calcific tendinopathy of shoulder: randomised double blinded multi-arm study. BMJ. 2023 Oct 11;383:e076447. doi: 10.1136/bmj-2023-076447. PMID 37821122